CLINICAL TRIAL: NCT03648853
Title: Effect of Location of Tetanic Stimuli on Photopethysmogram During General Anesthesia
Brief Title: Effect of Location of Tetanic Stimuli on Photoplethysmogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Pekka Talke, MD, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PT1801
Record Dates: First submitted 2018-08-24; First posted 2018-08-27 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Stress Reaction
Keywords: photoplethysmography; stress response
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- intervention (Experimental): all participants receive the same intervention
  Interventions: Device: Tetanic Stimulus

INTERVENTIONS:
Device: Tetanic Stimulus — 5 second 100 Hz 70 mA tetanic stimulus will be applied to three different locations in a random order

SUMMARY:
The effect of the location of tetanic stimulus on photoplethysmography signals will be studies in patients under general anesthesia.

DETAILED DESCRIPTION:
A 5 second 100 Hz 70 mA tetanic stimulus will be applied to three different locations in a random order in patients who are under general anesthesia. Tetanic stimuli are used routinely during general anesthesia to assess effectiveness of neuromuscular blockade. These tetanic stimuli are noxious stimuli that elicit a stress response which can be quantified using photoplethysmography. This study investigates if the magnitude of the tetanus induced stress response is dependent on the location of the tetanic stimulus as measured by photoplythysmography.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients general anesthesia able to consent in english

Exclusion Criteria:

* regional anesthesia unable to consent in english under 18 yrs of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talke P, Talke I. Effect of the Location of Tetanic Stimulation on Autonomic Responses: A Randomized Cross-Over Pilot Study. J Pain Res. 2024 Jan 9;17:209-217. doi: 10.2147/JPR.S443058. eCollection 2024. PMID 38223663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 surgical patients were recruited between 10/3/19/2018 and 11/30/2018. All subjects completed the study. Study was conducted in surgical patients under general anesthesia at UCSF
Groups:
- Intervention: All subjects received the same intervention
Period: Overall Study
Arm/Group | Intervention
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
photoplethysmagraph AC/DC values 60 seconds before each tetanic stimulus was considered as the basee [Mean (Standard Deviation); unit: arbitrary units] — photoplethysmographs (PPG) record transmitted infrared light through the finger. The PPG signal is recorded in arbitrary units (from A to D converter). The varying part of the signal (due to cardiac contractions) is called AC. The values from zero to the bottom of the varying part is called DC. In the study I used AC/DC*100. This ratio approximates the portion of the signal (in percent) that varies over time. A lower AC/DC is normally recorded when blood vessels are vasoconstricted. The baseline AC/DC in this study refers to the values immediately before intervention.
  arbitrary units | 5.4 (1.95)

OUTCOME MEASURES:

1. Primary Outcome: Photoplethysmography (PPG)
Description: Change in the PPG signal in response to tetanic stimulus. A tetanic stimulus will cause vasoconstriction which can be recorded as a decrease in PPG AC/DC. The outcome measure is the maximum decrease in AC/DC from baseline. Maximum decrease happens typically in 30-60 seconds after the stimulus. Thus, data was collected immediately before (baseline) and for 2 min after the stimulus. After the stimulus AC/DC values return to baseline in a few minutes. Baseline AC/DC measures a relative state of blood vessel tone. In anesthetized patients the AC/DC values can range from close to 0 to above 10. The higher the value, the more vasodilated the subject is.
Time Frame: 1-2 minutes
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Intervention
Number analyzed (Participants) | 12
arbitrary units | 3.3 (1.6)

ADVERSE EVENTS:
Time Frame: From beginning of general anesthesia till end of study data collection during general anesthesia which was approximately one hour.
Description: Tetanic stimulus (the only intervention of this study) has never been associated with adverse events. Tetanic stimulus is routinely used during general anesthesia to assess neuromusculer blockade.
Groups:
- Intervention: All subjects received the same intervention. There were no adverse effects
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT03648853/Prot_SAP_001.pdf